CLINICAL TRIAL: NCT01601353
Title: Evaluate the Use of Liposuction and Cell Separation Devices for Autologous Fat (Adipose) Derived Cells to Treat the Symptoms of Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tissue Genesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ED1001
Record Dates: First submitted 2012-05-09; First posted 2012-05-18 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Injection of adipose derived cells into penis
  Interventions: Device: Tissue Genesis Cell Isolation System
- Control (No Intervention): No intervention through 9 months

INTERVENTIONS:
Device: Tissue Genesis Cell Isolation System — Liposuction followed by injection of autologous adipose derived cells
  Arms: Treatment

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of adipose derived cells for the treatment of erectile dysfunction symptoms.

DETAILED DESCRIPTION:
This trial is being conducted to determine the safety and efficacy of injecting autologous adipose derived cells into the penis of men with erectile dysfunction. Subjects will be randomized into a treatment and control arm.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 40 - 70
2. Willing and able to provide written informed consent
3. Chronic, organic erectile dysfunction (ED), duration at least 0.5 years, with baseline International Index of Erectile Function - Erectile Function (IIEF-EF) score of < 26
4. Willing to complete questionnaires
5. Involved in a monogamous, heterosexual relationship for at least 3 months with both partners motivated to have or attempt sexual intercourse at least 4 times per month beginning two weeks after study treatment (subject reported)
6. Not interested or able to use oral PDE-5 inhibitor (PDE-5i) drug therapy, and willing to forgo these treatments for the first 6-month period following study treatment (in addition may include a minimum 4-week washout since last PDE-5i use prior to completion of the baseline erectile function assessments and study treatment)
7. Willing to limit alcohol intake and eliminate use of recreational drugs for sexual encounters
8. Willing to undergo a minor surgical procedure and injection
9. Abdominal area amenable to liposuction of at least 60-120 cc of adipose tissue based on Investigator examination
10. Mentally competent and able to understand all study requirements (based on investigator assessment)
11. Willing to be available for all baseline, treatment and follow-up examinations required by protocol
12. Willing to forego participation in any other study throughout the duration of this study unless receiving prior approval by Sponsor.

Exclusion Criteria:

1. Evidence of prostate cancer which requires additional radiotherapy or other adjuvant therapy
2. Previous pelvic or abdominal radiation therapy
3. Previous, concomitant or scheduled use of anti-androgen therapy
4. Untreated hypogonadism or low serum total testosterone (< 200 ng/dL)
5. Clinically evident penile anatomical deformities (e.g., Peyronie's disease) or history of priapism
6. Skin irritation, infection, wound, sore or disruption in the immediate areas of skin entry for abdominal liposuction or penile injection (including abdominal trauma and abdominal skin cancer (basal cell carcinoma, squamous cell carcinoma, and melanoma))
7. Use of any non-study treatment for erectile dysfunction within 4 weeks of study treatment and a lack of willingness to continue through 6 months after study treatment
8. Any previous penile implant or penile vascular surgery
9. Current or previous malignancy other than localized prostate cancer or nonabdominal, non-melanoma skin cancer (successfully treated or treatable by curative excision or other local curative therapy- abdominal skin cancer is exclusionary as indicated in criteria 6)
10. Uncontrolled hypertension or hypotension (systolic blood pressure > 170 or < 90 mm Hg, and diastolic blood pressure > 100 or < 50 mm Hg)
11. Reported unstable cardiovascular disease (e.g., unstable angina, myocardial infarction within past 6 months, cardiac failure or life-threatening arrhythmia, congestive heart failure) or symptomatic postural hypotension within 6 months before screening
12. Hemoglobin A1c > 8% within 8 weeks prior to study treatment
13. Current urinary tract or bladder infection
14. Drug, alcohol, or substance abuse reported within the last three years (subject reported)
15. Subject's sexual partner is < 18 years of age, nursing, or known to be pregnant at screening, or wishes to become pregnant during the study period, or has any gynecologic problems, major medical conditions, or other factors that would limit participation in sexual intercourse to less than 4 times per month (subject reported)
16. Weight less than 154 lbs/ 70 kg, or BMI ≥ 30
17. Unable to limit or avoid nonsteroidal anti-inflammatory drugs(NSAIDs) for 15 days prior to treatment (subject reported)
18. Bleeding or clotting disorder, use of anticoagulant therapy, or history of easy or excessive bruising
19. Lab values for Complete Blood Count(CBC), Prothrombin Time(PT)/Partial Thromboplastin Time(PTT)/International Normalized Ration(INR), liver function and creatinine falling outside the normal lab values (see section 5.3 for further detail)
20. Systemic autoimmune disorder
21. Significant active systemic or localized infection
22. Receiving immunosuppressant medications

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Adverse Events that occur during or after the procedure to measure safety and tolerability | 3 years
Erectile function | 6 months

SECONDARY OUTCOMES:
Continence | 3 years
Treatment assessment | 3 years
Erection hardness | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - San Diego Sexual Medicine, San Diego, California
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Khera M, Albersen M, Mulhall JP. Mesenchymal stem cell therapy for the treatment of erectile dysfunction. J Sex Med. 2015 May;12(5):1105-6. doi: 10.1111/jsm.12871. No abstract available. PMID 25974235